CLINICAL TRIAL: NCT00403130
Title: Phase II Open Label Study of Gemcitabine, Paclitaxel and Bevacizumab Combination as First Line Treatment for Metastatic Breast Cancer
Brief Title: Phase 2 Study of Gemzar, Taxol & Avastin Combination as 1st Line Treatment for Metastatic Breast Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: George Albert Fisher (Other)
Collaborators: Genentech, Inc. (Industry); Eli Lilly and Company (Industry)
Responsible Party: Sponsor-Investigator, George Albert Fisher, Associate Professor of Medicine, Stanford University
Organization: Stanford University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB-13761; 96052 (Other: Stanford University alternate IRB Number); BRSMTS0007 (Other: OnCore study number)
Record Dates: First submitted 2006-11-22; First posted 2006-11-23 (Estimated); Results first posted 2017-03-24 (Actual); Last update posted 2019-02-20 (Actual); Status verified 2019-01

CONDITIONS: Breast Cancer; Metastatic Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Gemcitabine; Paclitaxel; Bevacizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Phase II 3-drug regimen (Experimental): Gemcitabine + Paclitaxel + Bevacizumab
  Interventions: Drug: Gemcitabine; Drug: Paclitaxel; Drug: Bevacizumab

INTERVENTIONS:
Drug: Gemcitabine — Gemcitabine 1000 mg/m2 by IV infusion, days 1, 8, and 15 in 28-day cycles
  Other Names: Gemzar
Drug: Paclitaxel — Paclitaxel 80 mg/m2 by IV infusion, days 1, 8, and 15 in 28-day cycles
  Other Names: Taxol
Drug: Bevacizumab — Bevacizumab 10 mg/kg by IV infusion, days 1 and 15 in 28-day cycles
  Other Names: Avastin

SUMMARY:
Single-institution phase 2 trial investigating the efficacy of capecitabine, oxaliplatin and bevacizumab for patients with metastatic neuroendocrine tumors.

DETAILED DESCRIPTION:
This study will evaluate the time-to-progression (TTP) in patients with metastatic breast cancer, receiving 1st line therapy with bevacizumab in combination with paclitaxel and gemcitabine.

Secondary objectives will include response rates and overall survival (OS).

ELIGIBILITY:
INCLUSION CRITERIA

* Previously-untreated metastatic breast cancer. May have had prior chest wall irradiation or palliative radiation to bony sites for control of pain or fracture. These sites of disease, however, will not be considered as sites of measurable disease.
* Use of bisphosphonates will be permitted.
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1.
* Granulocyte count ≥ 1500/mm³
* Platelet count ≥ 100,000/mm³
* Hemoglobin ≥ 8.0 g/dL.
* Serum glutamic oxaloacetic transaminase (SGOT) / serum glutamic pyruvic transaminase (SGPT) ≤ 2.5 x the institutional upper limit of normal (ULN) if alkaline phosphatase is ≤ ULN or alkaline phosphatase may be up to 4 x ULN if transaminases are ≤ ULN.
* Total bilirubin within institutional limits of normal.
* Calculated creatinine clearance ≥ 30 mL/min using the formula: Ccr(mL/min) = [(140-age in years) X (wt in kg) X 0.85 (females)]/(72 x serum creatinine in mg/dL)
* ≥ 18 years of age.
* Prior anthracycline treatment in the adjuvant setting or prior chest wall radiation must have left ventricular ejection fraction (LVEF) within the institutional range of normal as assessed by pre-treatment multigated acquisition (MUGA) scan or echocardiogram (ECHO).
* All patients must give signed written informed consent.
* May have received adjuvant therapy as long as therapy complete > 12 months from study entry.
* Females of childbearing potential must have a negative pregnancy test taken ≤ 2 weeks prior to study enrollment, and must consent to the use of effective contraception during the study period and for 6months thereafter.

EXCLUSION CRITERIA

* Receiving hormonal therapy
* Prior treatment for metastatic disease with cytotoxic agents or inhibitors of epidermal growth factor receptor (EGFR)
* Her2NEU-positive breast cancers, by either immunohistochemistry (IHC) score 3+ or fluorescence in situ hybridization (FISH)
* Pregnant or lactating.
* Patients have had active malignancies other than breast cancer in the past 5 years with the exception of in situ carcinoma of the cervix or nonmelanomatous skin cancer.
* Active or unresolved infection.
* Pre-existing peripheral neuropathy > Grade 1.
* Prior history of severe hypersensitivity reaction to paclitaxel, gemcitabine, bevacizumab or drugs formulated with polysorbate 80.
* Current, recent (within 4 weeks of the first infusion of this study), or planned participation in an experimental drug study.
* Blood pressure of >150/100 mmHg
* Unstable angina
* New York Heart Association (NYHA) Grade II or greater congestive heart failure
* History of myocardial infarction within 6 months
* History of stroke within 6 months
* Clinically-significant peripheral vascular disease
* Evidence of bleeding diathesis or coagulopathy
* Presence of central nervous system or brain metastases
* Major surgical procedure, open biopsy, or significant traumatic injury within 28 days prior to Day 0, anticipation of need for major surgical procedure during the course of the study
* Minor surgical procedures, fine needle aspirations or core biopsies within 7 days prior to Day 0
* Urine protein:creatinine ratio ≥ 1.0 at screening
* History of abdominal fistula, gastrointestinal perforation, or intra-abdominal abscess within 6 months prior to Day 0
* Serious, non-healing wound, ulcer, or bone fracture
* Inability to comply with study and/or follow-up procedures

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2006-02; Primary Completion 2010-09 (Actual); Study Completion 2012-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: George A Fisher, MD, PhD, Principal Investigator — Stanford University
Locations (1):
- Stanford University School of Medicine, Stanford, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Guardino A, et al. "Phase II Trial with Gemcitabine, Paclitaxel and Bevacizumab for the First Line Treatment of Metastatic Breast Cancer." Cancer Res. 2009;69(24_suppl)abs6089.

RESULTS

PARTICIPANT FLOW:
Groups:
- Gemcitabine + Paclitaxel + Bevacizumab: * Gemcitabine 1000 mg/m2 by IV infusion, days 1, 8, and 15 in 28-day cycles
  * Paclitaxel 80 mg/m2 by IV infusion, days 1, 8, and 15 in 28-day cycles
  * Bevacizumab 10 mg/kg by IV infusion, days 1 and 15 in 28-day cycles
Period: 2 Years From Start of Treatment
Arm/Group | Gemcitabine + Paclitaxel + Bevacizumab
Started | 31
Completed | 26
Not Completed | 5
Not completed — Not Eligible | 3
Not completed — Lost to Follow up | 1
Not completed — Withdrawal by Subject | 1
Period: Survival Follow-up up to 6 Years
Arm/Group | Gemcitabine + Paclitaxel + Bevacizumab
Started | 26
Completed | 16
Not Completed | 10
Not completed — Lost to Follow-up | 10

BASELINE CHARACTERISTICS:
Arm/Group | Gemcitabine + Paclitaxel + Bevacizumab
Number analyzed (Participants) | 31
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 24
  >=65 years | 7
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 31
  Male | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 5
  Not Hispanic or Latino | 26
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 5
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 2
  White | 21
  More than one race | 1
  Unknown or Not Reported | 2

OUTCOME MEASURES:

1. Primary Outcome: Time-to-Progression (TTP)
Description: Time-to-Progression (TTP) was assessed as the time from start of treatment to progression, as observed on radiographic scans and assessed per the Response Evaluation Criteria in Solid Tumors (RECIST) v1.1 criteria for progressive disease (ie, a 5-mm absolute increase of the sum of the longest diameters of the target lesions in addition to a 20% increase in the sum of the target lesions)
Time Frame: 2 years
Population: Disease progression was documented for 9 participants.
Measure: Median (Standard Deviation); unit: months
Groups:
- Bevacizumab + Gemcitabine + Paclitaxel: * Gemcitabine 1000 mg/m2 by IV infusion, days 1, 8, and 15 in 28-day cycles
  * Paclitaxel 80 mg/m2 by IV infusion, days 1, 8, and 15 in 28-day cycles
  * Bevacizumab 10 mg/kg by IV infusion, days 1 and 15 in 28-day cycles
Arm/Group | Bevacizumab + Gemcitabine + Paclitaxel
Number analyzed (Participants) | 9
months | 8.9 (5.9)

2. Secondary Outcome: Response Rates
Description: The best overall response was recorded for each participant from randomization until disease progression/recurrence, using any increase from the smallest measurements recorded since randomization as the indicator of Progressive Disease (PD).
  Overall response was determined on the basis of response at the target and non-target lesions, and the appearance of new lesions, as follows.
  Target Nontarget New Lesions Overall Response
  * Complete Complete None Overall Complete Response
  * Complete Incomplete response/ None Overall Partial Response Stable Disease (SD)
  * Partial Not PD None Overall Partial Response
  * SD Not PD None Overall Stable Disease
  * PD Any Yes/No Overall PD
  * Any PD Yes/No Overall PD
  * Any Any Yes Overall PD
  Overall Response Rate (ORR) was assessed as the sum of the Complete Response (CR) rate and the Partial Response (PR) rate.
Time Frame: 24 weeks
Population: Although 24 participants completed treatment, only 13 were evaluable for treatment effect.
Measure: Count of Participants; unit: Participants
Arm/Group | Bevacizumab + Gemcitabine + Paclitaxel
Number analyzed (Participants) | 13
Participants
  Complete Response (CR) | 1
  Partial Response (PR) | 4
  Stable Disease (SD) | 1
  Progressive Disease (PD) | 7
  Overall Response Rate (ORR) | 5

3. Secondary Outcome: Overall Survival (OS), Confirmed
Description: Overall Survival (OS) as determined by confirmed date of death. Participants without documentation as either alive or deceased as of 6 years from the start of treatment were considered lost-to-follow-up.
Time Frame: 6 years
Measure: Median (Full Range); unit: months
Arm/Group | Bevacizumab + Gemcitabine + Paclitaxel
Number analyzed (Participants) | 16
months | 33.7 [13.8 to 66.9]

4. Secondary Outcome: Overall Survival (OS), All Participants
Description: Overall Survival (OS), based on date of death or last known date alive
Time Frame: 6 years
Measure: Median (Full Range); unit: months
Arm/Group | Bevacizumab + Gemcitabine + Paclitaxel
Number analyzed (Participants) | 26
months | 14.8 [5.0 to 66.9]

ADVERSE EVENTS:
Time Frame: 2 years
Arm/Group | Gemcitabine + Paclitaxel + Bevacizumab
Serious Adverse Events (participants affected / at risk) | 18/26
Other Adverse Events (participants affected / at risk) | 26/28
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Gemcitabine + Paclitaxel + Bevacizumab (N=26)
Thrombocytopenia (Blood and lymphatic system disorders) | 4 (8)
Weakness (General disorders) | 1 (1)
Acute Renal failure (Renal and urinary disorders) | 1 (1)
Aspartate Aminotransferase (Metabolism and nutrition disorders) | 1 (1) — serum glutamic oxaloacetic transaminase
Peripheral arterial ischemia (Cardiac disorders) | 1 (1)
Febrile neutropenia (Infections and infestations) | 1 (1)
Syncope (Nervous system disorders) | 1 (1)
Thrombosis (Cardiac disorders) | 1 (1) — Embolism
Neutropenia (Blood and lymphatic system disorders) | 3 (4)
Epitasis (Blood and lymphatic system disorders) | 1 (1)
Pain (General disorders) | 2 (2) — Includes: underneath breast, amputation area
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Gemcitabine + Paclitaxel + Bevacizumab (N=28)
Pain (General disorders) | 4 (4)
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 3 (3)
Shortness of breath (Respiratory, thoracic and mediastinal disorders) | 1 (1) — Mild
Alanine Aminotransferase, serum glutamic pyruvic transaminase (Blood and lymphatic system disorders) | 3 (6)
Aspartate Aminotransferase, serum glutamic oxaloacetic transaminase (Blood and lymphatic system disorders) | 3 (4)
Febrile neutropenia (Infections and infestations) | 6 (10)
Hypoglycemia (Blood and lymphatic system disorders) | 1 (1)
Thrombocytopenia (Blood and lymphatic system disorders) | 7 (10)
Neutropenia (Infections and infestations) | 11 (20)
Scalp folliculitis (Infections and infestations) | 1 (1)
Infection with normal absolute neutrophil count (Infections and infestations) | 1 (1)
Neutrophils/granulocytes (Blood and lymphatic system disorders) | 2 (6)
Hypertension (Blood and lymphatic system disorders) | 3 (3)
Proteinuria (Renal and urinary disorders) | 1 (1)
Leukopenia (Blood and lymphatic system disorders) | 5 (10)
Anorexia (Gastrointestinal disorders) | 1 (1)
Constipation (Gastrointestinal disorders) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 2 (2)
Dysphagia (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1)
Hypokalemia (Blood and lymphatic system disorders) | 1 (1)
Neuropathy (Nervous system disorders) | 1 (1)
Infection (Skin and subcutaneous tissue disorders) | 1 (1) — Cellulitis
Hypoalbuminemia (Blood and lymphatic system disorders) | 2 (2)
Anemia (Blood and lymphatic system disorders) | 2 (2)
Congestion (General disorders) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Epistaxis (Blood and lymphatic system disorders) | 3 (3)
Erythematous (Skin and subcutaneous tissue disorders) | 1 (1)
Fatigue (General disorders) | 3 (3)
Alopecia (Skin and subcutaneous tissue disorders) | 1 (2)
Headache (Nervous system disorders) | 4 (5)
Heartburn (Cardiac disorders) | 1 (1)
Urinary tract infection (Infections and infestations) | 2 (2)
Cellulitis (Skin and subcutaneous tissue disorders) | 2 (2)
Upper respiratory infection (Infections and infestations) | 2 (2)
Gingivitis (Infections and infestations) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 1 (1)
Irregular menses (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Shortness of breath (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Nail changes (Skin and subcutaneous tissue disorders) | 1 (1)
Peripheral neuropathy (Nervous system disorders) | 3 (4)
Proteinuria (Renal and urinary disorders) | 2 (3)
Thrombosis (Blood and lymphatic system disorders) | 2 (2) — embolism

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No